CLINICAL TRIAL: NCT05760625
Title: Gender Differences and Features of the Clinical Course of Primary Headaches
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Tashkent Medical Academy (Other)
Responsible Party: Principal Investigator, Bahtigul Holmuratova, Dr. Bahtigul, Tashkent Medical Academy
Other Study IDs: 616.857-036:616.831:615.21
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Primary Headache Disorder
Keywords: migraine; pain; attack; BDNF; neurotrophins
MeSH Terms: conditions — Headache Disorders, Primary; Migraine Disorders; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Migraine: In migraineurs, venous blood samples will be collected twice: outside and during migraine attacks prior to pain medication. Analysis of BDNF performed using enzyme-linked immunosorbent assay technique.
  Interventions: Diagnostic Test: analysis BDNF
- Tension type of headache: In patients with tension-type headache (outside attack) and healthy controls, one single blood sample will take. Analysis of BDNF performed using enzyme-linked immunosorbent assay technique.
  Interventions: Diagnostic Test: analysis BDNF
- Cluster headache: In cluster headache patients serum samples will be collected in and outside cluster bout. Analysis of BDNF performed using enzyme-linked immunosorbent assay technique.
  Interventions: Diagnostic Test: analysis BDNF

INTERVENTIONS:
Diagnostic Test: analysis BDNF — We analysed consentration of BDNF in venous blood of patient with primary headache

SUMMARY:
The pathophysiological mechanisms that underlie primary headache disorders, such as migraine and cluster headache (CH), are complex and not yet fully clarified. While there is today little doubt that activation of the trigeminovascular system (TGVS) is responsible for the headache pain, the primary mechanisms, probably centrally mediated, leading to its activation and the generation of pain are still largely obscure. The trigeminal system is supposed to play a central role not only in migraine but also in cluster headache pathology. In vitro studies have demonstrated the expression of BDNF in trigeminal ganglion neurons. BDNF release is induced by trigeminal stimulation and nociceptive inputs. BDNF is a member of the neurotrophin family and has been recognized as an important modulator of nociceptive pathways. Interestingly, BDNF is co-expressed with CGRP in trigeminal ganglion neurons. CGRP is one of the key molecules in migraine and cluster headache pathogenesis. BDNF is an important marker of neuronal plasticity. It has also been associated with pain processing. Increased BDNF levels are observed in chronic pain syndromes. In order to understand the role of BDNF associated with other factors such as gender on headache attacks we aimed to determine whether migraine and cluster headache is correlated with brain derived neurotrophic factor (BDNF) level, gender and age.

DETAILED DESCRIPTION:
Patients will recruite among those attending the Clinic of Tashkent Medical Academy, Uzbekistan. Three groups of headache patients will be enrolled in this prospective study: patients with episodic migraine with and without aura, episodic cluster headache, and frequent episodic tension-type headache according to the current criteria of the International Headache Society. In migraineurs, venous blood samples will be collected twice: outside and during migraine attacks prior to pain medication. In cluster headache patients serum samples will be collected in and outside cluster bout. Analysis of BDNF will performed using enzyme-linked immunosorbent assay technique. In patients with tension-type headache (outside attack) and healthy controls, one single blood sample will take.Patients with a history of cardiovascular disease, major depression, hypertension, drug or alcohol abuse, or other apparent diseases will be excluded from the study. The research will comprise 120 patients (males and females) suffering from primary headache. At the moment we started collecting patients.

ELIGIBILITY:
Inclusion Criteria:

* Migraine patients were included if they suffered from at least one, but no more than eight migraine attacks per month, and had not taken any pain medication including non-steroidal anti inflammatory drugs (NSAIDs), triptans or opioids 48 h prior to blood sample collection and if phone contact was possible 3 days after blood sampling.

Exclusion Criteria:

* Patients were not included if they had a history of cardio or cerebrovascular disease, diabetes, cancer, severe renal or hepatic disease. Patients with more than one diagnosis of a primary headache, i.e. coexistent migraine and tension-type headache, were excluded from study participation. Pregnancy and breastfeeding were additional exclusion criteria.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients, males and females, were included if they consented to study participation, and were aged between 18 and 45 years
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-12-10 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2023-03-21 (Estimated)

PRIMARY OUTCOMES:
Gender differences and features of the clinical course of primary headaches | 2 years
  Increasing of BDNF during headache attacks in women were more than men

CONTACTS AND LOCATIONS:
Overall Officials: Bahtigul Holmuratova, PhD student, Study Chair — Tashkent Medical Academy
Locations (1):
- Tashkent Medical Academy, Tashkent, Olmazor District, Uzbekistan

IPD SHARING:
Plan to Share IPD: No
The pathophysiological mechanisms that underlie primary headache disorders, such as migraine and cluster headache (CH), are complex and not yet fully clarified. While there is today little doubt that activation of the trigeminovascular system (TGVS) is responsible for the headache pain, the primary mechanisms, probably centrally mediated, leading to its activation and the generation of pain are still largely obscure. The trigeminal system is supposed to play a central role not only in migraine but also in cluster headache pathology. In vitro studies have demonstrated the expression of BDNF in trigeminal ganglion neurons. BDNF release is induced by trigeminal stimulation and nociceptive inputs.